CLINICAL TRIAL: NCT01862796
Title: Is Non-Adherence Unique to Weight-Loss? Predictors of Adherence to a Heart-Healthy Diet in Lean vs. Obese Individuals
Brief Title: Predicting Adherence to a Heart-Healthy Diet in Lean and Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 999913096; 13-DK-N096 (Other: NIDDK/NIH)
Record Dates: First submitted 2013-05-23; First posted 2013-05-24 (Estimated); Results first posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2018-05-22

CONDITIONS: Obesity; Overweight
Keywords: Food Intake; Weight Loss; Compliance
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Patient Compliance

ARMS (3):
- Obese underfeeding (UF) (Experimental): Obese randomized to received a 35% calorie reduced diet
  Interventions: Behavioral: Underfeeding diet
- Obese weight maintaining (WMEN) (Experimental): Randomized to receive a weight-maintaining diet
  Interventions: Behavioral: Weight maintaining diet
- Lean weight maintaining (WMEN) (Experimental): Normal weight individuals receiving a weight-maintaining energy needs diet
  Interventions: Behavioral: Weight maintaining diet

INTERVENTIONS:
Behavioral: Underfeeding diet — Heart healthy diet with 35% reduced calories
  Other Names: UF
  Arms: Obese underfeeding (UF)
Behavioral: Weight maintaining diet — Heart healthy weight-maintaining diet
  Other Names: WMEN
  Arms: Lean weight maintaining (WMEN); Obese weight maintaining (WMEN)

SUMMARY:
Background:

- Sticking to a diet plan can be difficult, but is important for many different health reasons. Some people seem to have a harder time following and sticking to a diet plan than others. It is not clear whether people of different weights (lean or obese) might have differences in the way they adhere to diet plans. Researchers want to study three different groups of people based on their body mass index (BMI), which measures people based on their weight and height. The study will place the participants on a 6-week diet and see how well they follow the diet. The information from this study may help develop better weight-loss plans and healthy diet ideas.

Objectives:

* To understand what factors affect adherence to a diet plan.
* To collect information for future studies that may improve people's ability to stick to diets.

Eligibility:

- Individuals at least 18 years of age who are lean (BMI between 18.5 and 25) or obese (BMI greater than 30).

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. They will have a full-body scan to measure fat and muscle. They will also answer questions on eating behaviors, mood, and desire to change eating patterns.
* Participants will be separated into three groups. Each group will have a different diet. The lean group will have a heart-healthy diet designed to maintain the same weight. One of the obese groups will also have a heart-healthy diet designed to maintain the same weight. The other obese group will have a heart-healthy weight loss diet. In all groups, all food will be provided by the study doctors. Participants should not eat any food other than that provided for the study.
* Everyone will start with a 1-week food testing period to find the right number of calories for each group. After this first week, participants will attend one diet counseling session per week and will be contacted randomly once a week to check on the foods they have had in the past 24 hours. Participants will complete daily food diaries on paper as well as daily food records using a smart phone.
* Participants will come to the clinic twice a week to pick up the diet food. On one of those days, they will also have their counseling session.
* The study will last for 6 weeks. At the final study visit, participants will repeat the tests from the screening study.

DETAILED DESCRIPTION:
Adherence, or "sticking to your diet" is important for successful initial weight loss and keeping off the weight over the long term (1). While early behavioral and dietary adherence have been associated with greater weight loss, sticking to a diet plan is difficult. It is not clear if adherence to any diet plan (even one which does not produce weight loss) is hard or whether people who are overweight have more difficulty with adhering to diet plans compared to people who are relatively lean.

The main aim of this study is to evaluate dietary adherence in 3 groups of individuals participating in a 6-week heart-healthy dietary intervention program. Two groups [1 (BMI < 25 kg/m(2)) and 2. Obese (BMI greater than or equal to 30 kg/m(2))] will receive a heart-healthy diet designed to maintain their weight, and the third group [3. Obese] will be given a heart-healthy diet that is 35% less than their daily calorie needs to lose weight. Participants will attend one counseling session per week and will be contacted randomly 1x/week by study staff for completion of a 24-hour dietary recall. They will complete daily food diaries and daily records using smart-phones. Prior to starting the assigned heart-healthy dietary intervention, participants will complete questionnaires that include questions about how motivated they are to follow a diet, lose weight, and change eating patterns. These findings may help us understand what factors affect adherence, and help us design weight loss studies that improve people's ability to stick to diet interventions.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. BMI

   * BMI greater than or equal to 30 kg/m(2) for the obese WMEN and UF groups but body weight less than 350 pounds to accommodate the DXA scanner
   * BMI less than or equal to 25 kg/m(2) (and BMI greater than or equal to 18.5 kg/m(2)) for the lean WMEN group
2. Age greater than or equal to 18 years. Minors under the age of 18 will be excluded because growth and pubertal issues are significant parameters that could affect our outcomes and also because the time requirements of the study are such that they would interfere with school schedules. Participants must be healthy, as determined by medical history, physical examination, and laboratory tests.
3. Weight stable (plus or minus 2 percent) for last 3 months

EXCLUSION CRITERIA:

Candidates will be screened by phone to exclude those with BMI greater than or equal to 26 kg/m(2) and BMI less than or equal to 29 kg/m(2), significant health problems, including cancer, hypertension, diabetes, current and past 3-month use of certain prescribed medications, especially those that could affect body weight, such as antidepressants and stimulants as well as smoking, or excess alcohol (greater than 3 drinks/d). Women must not be pregnant or lactating, and be at least 1 year postpartum. Candidates with a history of psychotic disorder or hospitalization for psychiatric illness within the past 1 year will not be eligible. They will need to be weight stable for the past 3 months (plus or minus 2 percent) and cannot be in treatment for obesity or currently receiving psychotherapy. Individuals who meet criteria according to the phone screen will be invited to come to the unit for a screening visit and their screening sheets are placed in a locked filing cabinet. Forms from potential volunteers who are ineligible are shredded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05-31; Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marci Gluck, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Fappa E, Yannakoulia M, Pitsavos C, Skoumas I, Valourdou S, Stefanadis C. Lifestyle intervention in the management of metabolic syndrome: could we improve adherence issues? Nutrition. 2008 Mar;24(3):286-91. doi: 10.1016/j.nut.2007.11.008. Epub 2008 Jan 16. PMID 18201869
- [Background] Flegal KM, Graubard BI, Williamson DF, Gail MH. Weight-associated deaths in the United States. J Womens Health (Larchmt). 2007 Nov;16(9):1368-70. doi: 10.1089/jwh.2007.0547. No abstract available. PMID 18001195
- [Background] Kassirer JP, Angell M. Losing weight--an ill-fated New Year's resolution. N Engl J Med. 1998 Jan 1;338(1):52-4. doi: 10.1056/NEJM199801013380109. No abstract available. PMID 9414332
- [Derived] Stinson EJ, Piaggi P, Votruba SB, Venti C, Lovato-Morales B, Engel S, Krakoff J, Gluck ME. Is Dietary Nonadherence Unique to Obesity and Weight Loss? Results From a Randomized Clinical Trial. Obesity (Silver Spring). 2020 Nov;28(11):2020-2027. doi: 10.1002/oby.23008. PMID 32808484

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 100 participants were assessed for eligibility, 30 were ineligible and 9 did not complete the run-in phase. Sixty-one were assigned to groups.
Period: Overall Study
Arm/Group | Obese Underfeeding (UF) | Obese Weight Maintaining (WMEN) | Lean Weight Maintaining (WMEN)
Started | 19 | 18 | 24
Completed | 19 | 18 | 23
Not Completed | 0 | 0 | 1
Not completed — Prohibited medications | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese Underfeeding (UF) | Obese Weight Maintaining (WMEN) | Lean Weight Maintaining (WMEN) | Total
Number analyzed (Participants) | 19 | 18 | 23 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (16.8) | 49.8 (13.1) | 49.7 (12.5) | 48.3 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 14 | 37
  Male | 9 | 5 | 9 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethniticy: American Indian or Alaskan Native | 7 | 8 | 1 | 16
  Race/Ethniticy: Asian | 0 | 0 | 1 | 1
  Race/Ethniticy: Native Hawaiian of Pacific Islander | 1 | 0 | 0 | 1
  Race/Ethniticy: Black or African American | 0 | 2 | 3 | 5
  Race/Ethniticy: Hispanic/Latino | 2 | 5 | 1 | 8
  Race/Ethniticy: Caucasian | 9 | 3 | 17 | 29
Region of Enrollment [Number; unit: participants]
  United States | 19 | 18 | 23 | 60
Weight, kg [Mean (Standard Deviation); unit: kg] | 111.0 (29.1) | 88.1 (15.3) | 63.9 (8.0) | 86.1 (27.3)
Height, cm [Mean (Standard Deviation); unit: cm] | 170.5 (10.4) | 161.7 (9.4) | 166.9 (8.6) | 166.5 (9.9)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 38.0 (8.7) | 33.5 (4.0) | 22.9 (1.8) | 30.9 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Adherence Score
Description: An adherence score is calculated each week by summing 7 measurements of adherence and dividing by 21, the maximum score, with range from 0 (no adherence) to 1 (perfectly adherent). For each of the 7 measures a higher score means better adherence: [1] Attendance (0-2), [2] Food diaries (0-3), [3] 24-hour food recall via interview (0-3), [4] computer survey (0-3), [5] 24-hour food recall via interview (0-3), [6] Ecological momentary assessment (0-6), and [7] On time arrival for session (0-1). The final score is calculated as the average of the six weekly scores.
Time Frame: Average over 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Obese Underfeeding (UF) | Obese Weight Maintaining (WMEN) | Lean Weight Maintaining (WMEN)
Number analyzed (Participants) | 19 | 18 | 23
score on a scale | 0.57 (0.17) | 0.54 (0.18) | 0.59 (0.10)

2. Secondary Outcome: Change in Weight From Baseline to 6 Weeks
Description: Weight loss from baseline, calculated as weight at 6 weeks - weight at baseline
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Obese Underfeeding (UF) | Obese Weight Maintaining (WMEN) | Lean Weight Maintaining (WMEN)
Number analyzed (Participants) | 19 | 18 | 23
kg | -3.14 (2.76) | -1.64 (2.41) | -0.54 (1.53)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Obese Underfeeding (UF) | Obese Weight Maintaining (WMEN) | Lean Weight Maintaining (WMEN)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/23
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT01862796/Prot_SAP_000.pdf